CLINICAL TRIAL: NCT06026709
Title: Effectiveness and Cost-effectiveness of an Integrated Digital Psychological Intervention (EmoEase) in Chinese COPD Patients: Study Protocol of a Randomized Controlled Trial
Brief Title: Effectiveness and Cost-effectiveness of Digital Psychological Intervention (EmoEase) in Chinese COPD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Simiao Chen, professor, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CAMS&PUMC-IEC-2023-018
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Depression; Anxiety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- usual care + EmoEase group (Experimental): EmoEase, the digital intervention, will be delivered through a WeChat Mini Program. It will integrate two main pieces of training for anxiety and depression. We will develop the training mainly based on CBT.
  Interventions: Behavioral: EmoEase
- usual care (No Intervention): We will distribute informational pamphlets to participants in both the intervention and control groups, which will include guidance on the following aspects of self-management of COPD:23
  1. Concise overview of COPD, encompassing its definition, prevalent risk factors, commonly observed symptoms, and disease progression;
  2. Minimizing exposure to high-risk factors, such as tobacco/smoke exposure, air pollutants, household cooking emissions, and respiratory infections; .......
  (10) Receiving vaccinations for influenza and streptococcus pneumoniae.

INTERVENTIONS:
Behavioral: EmoEase — The online intervention"EmoEase" integrates two distinct trainings for anxiety and depression. Each training includes approximately twenty 10-minute sessions, and each are centered around different themes. These two trainings will be delivered through a WeChat Mini Program.
  Arms: usual care + EmoEase group

SUMMARY:
Background Mental health issues are common and often overlooked in COPD patients. Digital psychological interventions might help, but their effectiveness in Chinese COPD patients hasn't been studied. This study aims to develop and evaluate EmoEase, a digital psychological intervention, for its effectiveness and cost-effectiveness in improving mental wellbeing in Chinese COPD patients.

Methods This multicenter, two-arm, randomized controlled trial (RCT) will enroll at least 420 COPD patients over 35 years old. Participants will receive either usual care (control group) or usual care plus EmoEase (intervention group). Assessments will occur at baseline (T0), 4 weeks (T1), 8 weeks (T2), and 16 weeks (T3). Participants will complete questionnaires and undergo physical measurements. The primary outcome will be mental wellbeing measured by the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS). Secondary outcomes will assess mental and physical health, COPD symptoms, health risk behaviors, socioeconomic factors, and healthcare use and costs. Analyses will use an intention-to-treat approach.

Discussion This is the first RCT to evaluate EmoEase for COPD patients. If effective and cost-effective, EmoEase could be scaled up to provide mental health support to COPD patients in China.

DETAILED DESCRIPTION:
Background Mental health problems in chronic obstructive pulmonary disease (COPD) patients are common and frequently neglected. Digital psychological interventions may reduce mental health problems, but their effectiveness has not been evaluated in the Chinese COPD population. In this study, we will develop an integrated digital psychological intervention (EmoEase) and evaluate its effectiveness and cost-effectiveness in enhancing the mental wellbeing of COPD patients in China.

Methods This study is a multicenter, two-arm, randomized controlled trial (RCT) with a parallel-group design to enroll at least 420 COPD patients with age over 35 years. Participants will be assigned to receive either usual care (control group) or usual care + EmoEase (intervention group). Assessments will take place at baseline (T0) and 4 weeks (T1), 8 weeks (T2), and 16 weeks (T3) after baseline, and participants will be asked to complete questionnaires and have physical measurements taken. The primary outcome measure will assess mental wellbeing using the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS). Secondary outcome measures will assess mental health, physical health, COPD symptoms, health risk behaviors, socioeconomic indicators, and healthcare utilization and expenditure. Analyses will utilize an intention-to-treat approach.

Discussion This is the first RCT to examine the value of EmoEase, a novel digital psychological intervention for COPD patients. If this intervention is effective and cost-effective, it could be rapidly scaled up to provide mental health care for COPD patients in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35 years or older;
2. Post-bronchodilator FEV1/FVC ≤70% or confirmed COPD patients;
3. Literate and able to type;
4. Have a smartphone;
5. Be proficient in using the WeChat applet;
6. Willingness to self-help iCBT sessions for 8 weeks, 10-20 minutes of practice per session, roughly 1 hour per week, time and place flexible;
7. Receive three follow-up visits within four months (2 offline, 1 online) and complete a physical exam and online questionnaire; and
8. Willingness to provide the hospital with their usual cell phone number.

Exclusion Criteria:

1. Patients with a physician diagnosis of asthma or asthma-COPD overlap syndrome;
2. Patients hospitalized for COPD within the previous one year;
3. Having severe cognitive dysfunction and being unable to communicate;
4. Severely ill with less than 12-month life expectancy.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) | at baseline (T0), 4 weeks (T1), 8 weeks (T2), and 16 weeks (T3) after baseline
  Patients' mental wellbeing at baseline, and each follow-up is assessed using the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS). The Chinese version of the scale shows good psychometric properties WEMWBS is a self-report measure comprising 14 short statements focusing on positive wellbeing. Each statement is rated on a 5-point Likert scale, resulting in scores ranging from 14 to 70 (a higher score indicates better mental wellbeing).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen S, Chen W, Li Y, Yu Y, Chen Q, Jiao L, Huang K, Tong X, Geldsetzer P, Bunker A, Fang X, Jing S, Liu Y, Li Y, He L, Wang C, Wang W, Zheng Z, Zhang S, Zhao J, Yang T, Barnighausen T, Wang C. Effectiveness and cost-effectiveness of an integrated digital psychological intervention (EmoEase) in Chinese chronic obstructive pulmonary disease patients: Study protocol of a randomized controlled trial. Digit Health. 2024 Oct 1;10:20552076241277650. doi: 10.1177/20552076241277650. eCollection 2024 Jan-Dec. PMID 39381816